CLINICAL TRIAL: NCT01498562
Title: Randomized Phase II Study of Gefitinib Plus Nimotuzumab Versus Gefitinib in Patients With Advanced Non-small Cell Lung Cancer: Dual-agent Molecular Targeting of EGFR (DATE)
Brief Title: Phase II Study of Gefitinib Plus Nimotuzumab Versus Gefitinib in Non-small Cell Lung Cancer
Acronym: DATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0662
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gefitinib plus Nimotuzumab (Experimental): Combination therapy group: Gefitinib(250mg daily) and Nimotuzumab (200mg weekly)
  Interventions: Drug: Gefitinib and Nimotuzumab
- Gefitinib alone (Active Comparator): Mono-therapy group: Gefitinib(250mg daily)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib and Nimotuzumab — Combination therapy group: Gefitinib(250mg daily) + Nimotuzumab (200mg weekly)
  Other Names: h-R3
  Arms: Gefitinib plus Nimotuzumab
Drug: Gefitinib — Mono-therapy group: Gefitinib(250mg daily)
  Other Names: Iressa
  Arms: Gefitinib alone

SUMMARY:
Combining nimotuzumab to gefitinib may not only potentiate cellular cytotoxicity, but may also assist in overcoming inherent or acquired resistance to gefitinib alone.

DETAILED DESCRIPTION:
Reversible EGFR tyrosine kinase inhibitors (TKI), such as gefitinib, were shown to be effective in patients with non-small cell lung cancer (NSCLC). However, patients almost invariably develop resistance to TKIs and have disease progression. Nimotuzumab is a humanized monoclonal antibody targeting the EGFR.

Combining nimotuzumab to gefitinib may not only potentiate cellular cytotoxicity, but may also assist in overcoming inherent or acquired resistance to gefitinib alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study specific procedures
* Unresectable non-small cell lung cancer
* ECOG performance status of 0 to 2
* Male or female; ≥ 20 years of age
* Subjects whose disease has progressed after platinum-based chemotherapy
* Subjects with measurable lesion

Exclusion Criteria:

* Inadequate organ functions
* Disease progression after 2 or more previous chemotherapy regimens
* Prior therapy with EGFR-tyrosine kinase inhibitor or Anti-EGFR Monoclonal Ab
* Any clinically significant gastrointestinal abnormalities
* Past medical history of interstitial lung disease
* Pregnant or lactating female

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate at 3 months | 3 months after randomization of last patient
  The progression-free survival rate at 3 months of the patients with no progression of disease or death due to any cause until 3 months is elapsed after being randomized.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 3 months after randomization of last patient
  Progression free survival (PFS) defined as the time from randomized date to the progression date or the preceded date of death date due to any cause.
Overall survival (OS) | 3 months after randomization of last patient
  Overall survival (OS) defined as the period from randomly assigned point of time to the date of death due to any cause.
Overall safety profile | 3 months after randomization of last patient
  Overall safety profile verified as relevance of adverse events and laboratory abnormality in the study and grades granted based on (USA National Cancer Center) Common Terminology Criteria for Adverse Events such as the type, frequency and severity (CTCAE), v4.0.
Objective response rate (ORR) | 3 months after randomization of last patient
  Overall objective response rate (ORR) is the best response rate stipulated as complete response (CR) or partial response (PR) (target lesion and tumor response defined according to RECIST guideline version 1.1) and identified as percentage of the confirmed patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Yonsei Cancer Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HR, Jang JS, Sun JM, Ahn MJ, Kim DW, Jung I, Lee KH, Kim JH, Lee DH, Kim SW, Cho BC. A randomized, phase II study of gefitinib alone versus nimotuzumab plus gefitinib after platinum-based chemotherapy in advanced non-small cell lung cancer (KCSG LU12-01). Oncotarget. 2017 Feb 28;8(9):15943-15951. doi: 10.18632/oncotarget.13056. PMID 27823977
- See also: PI site — http://www.iseverance.com/